CLINICAL TRIAL: NCT01427660
Title: Technologically Enhanced Community Health Worker (CHW) Delivery of Personalized Diabetes Information
Brief Title: iDecide.Decido: Diabetes Medication Decision Support Study
Acronym: iDecide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Mase, Project Manager, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R18HS019256-01 (AHRQ)
Record Dates: First submitted 2011-08-31; First posted 2011-09-01 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes, Type 2
Keywords: Diabetes; Decision Aid; AntiHyperglycemic Medication; Tailored health information; Medication information
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional CERSG Arm (Active Comparator): CHWs will provide and review with patients language-appropriate versions of the AHRQ consumer guides. CHWs will highlight key points on each page, review information on each medication and elicit and address questions. They will use the autonomy enhancing, motivational-interviewing based skills. As with the first arm, CHWs will schedule follow-up clinic appointments for participants who note a specific treatment change they would consider and will call participants two times after the session at three and six weeks to address additional questions and to follow up on any goals the participant set.
  Interventions: Behavioral: Community Health Worker Diabetes Education: Print media
- Web-Based Materials Arm (Experimental): Participants randomized to this arm will be scheduled within 3 weeks of enrollment to have a one-hour face-to-face session with a CHW who will deliver the ipad platform personally tailored diabetes medication decision aid. Participants will receive a printed tailored preference summary at the completion of this visit. If participants note a specific treatment change they would like to discuss with their providers, the CHW will facilitate scheduling a clinic visit within the next month. Finally, CHWs will call participants two times after the session at 3 and 6 weeks to assess if the participant has additional questions and to follow up on any treatment or other goals the participant set during their session.
  Interventions: Behavioral: CHW Diabetes Education: tailored web site

INTERVENTIONS:
Behavioral: Community Health Worker Diabetes Education: Print media — Providing information to patients about potential benefits, harms, costs, and burdens of medications and discussing patients' treatment preferences.
  Other Names: Print Materials Arm
  Arms: Traditional CERSG Arm
Behavioral: CHW Diabetes Education: tailored web site — Providing tailored and interactive information to patients about potential benefits, harms, costs, and burdens of medications and discussing patients' treatment preferences.
  Other Names: Tailored web based decision aid
  Arms: Web-Based Materials Arm

SUMMARY:
Two of AHRQ 's consumer-focused guides, "Pills for Type 2 Diabetes" and "Premixed Insulin for Type 2 Diabetes" could be of great use to underserved ethnic and racial minority adults. The presentation of content and delivery mechanisms of these Guides, however, needs to be modified to increase their use and impact among these difficult-to-reach populations.

To achieve this goal, a long-standing collaboration among African American and Latino community organizations, health care centers and systems, public health organizations, and academics (the REACH Detroit Partnership) is joining with leading experts in the development of personally and culturally tailored health decision aids (University of Michigan's Center for Health Communications Research [CHCR] and Center for Behavioral and Decision Sciences in Medicine [CBDSM]).

The investigators will develop and evaluate a computer tailored online diabetes medication decision aid that will enable community health workers (CHWs) to provide personalized patient education materials to underserved diabetic African American and Latino adults in Detroit, Michigan.

DETAILED DESCRIPTION:
The Specific Aims of this study are:

Aim 1: To use the information in the two diabetes medications consumer CERSGs to build an interactive, computer tailored diabetes medication guide that will enable patients to assess their treatment goals, personal preferences, and side-effect concerns and generate a personally tailored assessment of their current diabetes treatments with, as appropriate, options for improving their diabetes care;

Aim 2: To determine the extent to which this personally tailored diabetes medication guide compared with the print consumer guides reduces Latino and African American diabetes patients' decisional conflict, through improved knowledge of anti-hyperglycemic medications and satisfaction with information received.

Aim 3: To examine the computer tailored program's effects on participants' changes in medications (medication intensification), self-reported medication adherence and beliefs and A1C levels between baseline and follow-up compared to participants receiving the print consumer guides.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* stated concern about diabetes and diabetes treatment
* poor glycemic control
* over 21 years of age

Exclusion Criteria:

* blind, deaf, otherwise unable to use the telephone or visual resources
* pregnant
* currently enrolled in other REACH Detroit research study
* in hospice care
* current radiation or chemotherapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in decisional conflict | baseline and 3 month post intervention
  We will be measuring subjects' perceptions of: a) uncertainty in choosing options; b) modifiable factors contributing to uncertainty such as feeling uninformed, unclear about personal values and unsupported in decision making; and c) effective decision making such as feeling the choice is informed, values-based, likely to be implemented and expressing satisfaction with the choice.

SECONDARY OUTCOMES:
Medication adherence and intensification | baseline and 3 month post intervention
  Self-reported medication adherence will be assessed through three well-validated measures. We will assess changes in anti-hyperglycemic medication dosages and/or numbers of medications by patient report and medical record review.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Heisler, MD, Principal Investigator — University of Michigan Meidcal School; Ann Arbor VA Center for Clinical Management Research,
Locations (1):
- Community Health and Social Service (CHASS), Detroit, Michigan, United States

REFERENCES:
- [Derived] Heisler M, Choi H, Palmisano G, Mase R, Richardson C, Fagerlin A, Montori VM, Spencer M, An LC. Comparison of community health worker-led diabetes medication decision-making support for low-income Latino and African American adults with diabetes using e-health tools versus print materials: a randomized, controlled trial. Ann Intern Med. 2014 Nov 18;161(10 Suppl):S13-22. doi: 10.7326/M13-3012. PMID 25402398